CLINICAL TRIAL: NCT01130870
Title: Dose Response Curve - Sacral Nerve Stimulation for Faecal Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 002; 002
Record Dates: First submitted 2010-05-14; First posted 2010-05-26 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Fecal Incontinence
Keywords: Fecal incontinence; Sacral nerve stimulation; Quality of life; DR15.9 Incontinentia alva
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sensory threshold - Amplitude (Active Comparator): Stimulation amplitude set at sensory threshold.
  Interventions: Device: Sensory Threshold
- 25% below sensory threshold - Amplitude (Experimental): Stimulation amplitude 75% of sensory threshold.
  Interventions: Device: 75% of sensory threshold - Amplitude
- 50% below sensory threshold - Amplitude (Experimental): Stimulation with amplitude set 50% below sensory threshold
  Interventions: Device: 50% of sensory threshold - Amplitude

INTERVENTIONS:
Device: Sensory Threshold — Sacral nerve stimulation with amplitude (sensory threshold), Frequency 14 Hz and pulse width 210 mic.sec.
  Arms: Sensory threshold - Amplitude
Device: 75% of sensory threshold - Amplitude — Sacral nerve stimulation with amplitude (75% of sensory threshold), Frequency 14 Hz and pulse width 210 mic.sec.
  Arms: 25% below sensory threshold - Amplitude
Device: 50% of sensory threshold - Amplitude — Sacral nerve stimulation with amplitude (50% of sensory threshold), Frequency 14 Hz and pulse width 210 mic.sec.
  Arms: 50% below sensory threshold - Amplitude

SUMMARY:
The purpose of this study is to determine if subsensory stimulation (amplitude) will maintain same continence in patients treated with Sacral Nerve Stimulation (SNS) for faecal incontinence as stimulation with amplitude at sensory threshold.

DETAILED DESCRIPTION:
Faecal incontinence is a devastating condition with huge impact on quality of life. Sacral Nerve Stimulation (SNS) has since 1995 been a treatment option for patients not obtaining satisfactory continence result with standard non-surgical treatments. SNS is electrical stimulation of the sacral nerve root(s2,3 or 4). Stimulation of this nerve roots results in improved continence. The mechanism of action is at present not well described.

Standard the neuromodulator (pacemaker) stimulate with Frequency 14 Hz, pulse width 210 mic.sec. and amplitude set at sensory threshold. One study by SM. Koch et all confirms that subsensory stimulation can be effective. At present there is no doubled blinded study's to confirm this theory of effective sub sensory stimulation.

The aim of this study is to determine if subsensory stimulation will be as effective as stimulation with amplitude at sensory threshold. This will be investigated in 20 patients who have had at least a reduction in incontinence episodes or Wexner inc. score of 75 % between preimplantation and latest follow up. The patients will be randomized to three different amplitudes. 1: amplitude set at sensory threshold. 2: 75% of sensory threshold. 3: 50% of sensory threshold. The order of the three settings will be random and in a double blinded manner. The interval between these three pacemaker settings is four weeks. Patients serve as there own controls. Stimulation frequency (14 Hz) and pulse width (210 mic-sec) will remain fixed.

Evaluation will be by means of 4 week bowel habit diary and questionnaires (Wexner inc. score / St. Marks Score / Wexner constipation score / Altomares OD-score / IBS-score/ Rockwood FIQoL -score). All patients will be evaluated with anorectal measurements (sphincter strength and anorectal volume measurements) before any changes of stimulation amplitude.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Informed consent
* Idiopathic fecal incontinence or Fecal incontinence due to small sphincter defect(≤60 o)
* fecal incontinence after primary/secondary sphincter repair
* Permanent neuromodulator (medtronic InterStim / Interstim II) implanted for at least 12 weeks before entering the study.
* Reduction in fecal incontinence episodes of at least 75% between baseline and latest follow up.(Bowel diary card) or 75% reduction of Wexner Inc. score.
* Willing and competent to fill out diary cards

Exclusion Criteria:

* Colorectal/proctological surgery since IPG-implant
* Pregnancy
* Anorectal Pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Number of incontinence episodes Assess number of incontinence episodes. | Will be assessed every four weeks during a twelve-week period
  Assess number of incontinence episodes, by means of bowel habit diary. Four week bowel habit diary will be evaluated three times during the twelve-week protocol perioed.

SECONDARY OUTCOMES:
Assess changes in anorectal volume and pressure with different amplitude. | Will be assessed every four weeks during a twelve-week period
  Resting and maximal anal sphincter pressure will be measured with different amplitude settings. In total three evaluations will be made in the twelve week protocol perioed.
Assess Quality of life after decrease in stimulation amplitude. | Will be assessed every four weeks during a twelve-week period
  Quality of life will be recorded by means of Rockwood faecal incontinence quality of life score. A total of three evaluations will be made every fourth week in the twelve week protocol perioed.

CONTACTS AND LOCATIONS:
Locations (1):
- Anal Physiology Laboratory, Surgical Research Section 900, Aarhus University Hospital, Aarhus, Aarhus C, Denmark

REFERENCES:
- [Derived] Duelund-Jakobsen J, Buntzen S, Lundby L, Laurberg S. Sacral nerve stimulation at subsensory threshold does not compromise treatment efficacy: results from a randomized, blinded crossover study. Ann Surg. 2013 Feb;257(2):219-23. doi: 10.1097/SLA.0b013e318269d493. PMID 23001079